CLINICAL TRIAL: NCT01829698
Title: Evaluate the Efficacy And Safety Of TUDCA Compare UDCA In The Treatment Of Cholestatic Liver Disease-PBC by A Randomized,Double-Blind,Double Dummy,Parallel-Controlled,Multicenter Trial and The Consecutive Treatment By TUDCA
Brief Title: Efficacy and Safety Study of TUDCA Compare UDCA to Treatment Chronic Cholestatic Liver Disease-PBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Trendful Kangjian Medical Information Consulting Limited Company (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trendful-TAU-001; 2009L05707 (Other Grant/Funding Number: SFDA)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Cholestatic Liver Disease
Keywords: tudca PBC Cholestasis tauroursodeoxycholic acid taurolite
MeSH Terms: interventions — ursodoxicoltaurine; Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tauroursodeoxycholic (Experimental): tauroursodeoxycholic acid, 750mg , divided into three times, each time 250mg, oral administration, after meal
  Interventions: Drug: tauroursodeoxycholic
- ursodeoxycholic (Active Comparator): control arm: ursodeoxycholic acid, 750mg ,divided into three times, each time 250mg, oral administration, after meal
  Interventions: Drug: ursodeoxycholic acid

INTERVENTIONS:
Drug: tauroursodeoxycholic — Testing arm: tauroursodeoxycholic acid, 750mg , divided into three times, each time 250mg, oral administration, after meal
  Other Names: TUDCA; Taurolite
  Arms: tauroursodeoxycholic
Drug: ursodeoxycholic acid — ursodeoxycholic acid, 750mg ,divided into three times, each time 250mg, oral administration, after meal
  Other Names: UDCA; Ursofalk
  Arms: ursodeoxycholic

SUMMARY:
Though ursodeoxycholate acid (UDCA) is the well known effective therapy for PBC,clinical effectiveness of UDCA may be limited by its poor absorption and extensive biotransformation.The more hydrophillic bile acid tauroursodeoxycholate (TUDCA) is the active ingredients of UDCA,and has been approved by state food and drug administration in China for treatment of cholesterol stones.So it is necessary to verify the efficacy and safety of TUDCA in the treatment of adult primary biliary cirrhosis. In this randomized, double-blinded, double -dummy, parallel-controlled and multicenter clinical trial, we detect the proportion of patients who had AKP decline more than 25% as the primary outcome;decline of ALP,total bilirubin, GGT,ALT and AST as secondary outcomes after patients were treated with TUDCA or UDCA for 24 weeks.

DETAILED DESCRIPTION:
This is a double-blind, randomized, parallel controlled, multicenter, clinical trial. Subjects inclusion by randomization after passing the screening, continuous administration the test drug (Taurolite) or control drug (Ursofalk) treatment for 24 weeks. Compare the safety and efficacy of Taurolite vs Ursofalk.

At the end of the double-blind period，enroll 100 subjects from both two group randomly ,for a consecutive treatment use TUDCA up to 24 weeks. Further evaluate the efficacy and safety of tauroursodeoxycholic acid (TUDCA) in the treatment of adult primary biliary cirrhosis (PBC) for a long time up to one year. Also evaluate the regimen's efficacy and safety that udca take placed by TUDCA in the treatment of adult primary biliary cirrhosis (PBC) for the patients who use udca treatment for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 1 Ages Eligible for Study: 18 Years to 70 Years

  2 Alkaline phosphatase (ALP) ≥ 2 times the Upper Limits of Normal (ULN);

  3 Anti mitochondrial antibody (AMA) positive and / or anti-mitochondrial antibody subtype M2 (AMA-M2) positive; if the AMA and AMA-M2 were negative, need liver biopsy confirmed pathological changes in PBC.

Exclusion Criteria:

* 1．in the 3 months before screening received UDCA, hormones, immunosuppressive therapy;

  2．with extrahepatic biliary obstruction;

  3．accompanied by hepatitis B virus (HBV) and hepatitis C virus (HCV) infection;

  4．laboratory screening examination :
  1. hemoglobin (HB): male< 11 g/dL, female <10 g/dL < g/dL;
  2. the total white blood cell (WBC) count < 3000/mm3;
  3. the absolute neutrophil count (ANC) <1500/mm3;
  4. platelet (PLT) count <50000/mm3;
  5. serum albumin <3.3g/dL;
  6. alanine aminotransferase (ALT) ≥ 10 ULN and / or aspartate aminotransferase (AST) ≥ 10ULN;
  7. ALT ≥ 5 ULN and / or AST ≥ 5 ULN with immunoglobulin G (IgG) ≥ 2ULN;
  8. total bilirubin (T-Bil) ≥ 4 ULN;
  9. prothrombin time (PT) prolonged ≥ 3 seconds (limit reference value based on) or PTA ≤ 60%;
  10. the serum creatinine (Cr) ≥ 1.5ULN.

  5．patients with esophageal variceal or bleeding, ascites, hepatic encephalopathy or other evidence of hepatic decompensation;

  6．diagnosed with liver cancer, suspected to have liver cancer, AFP > 100ng/ml. As the AFP in 2 times the upper limit of normal to 100ng/ml, need re-check in 2 weeks, if their AFP > 100ng/ml can not be included

  7．body mass index >28 (Kg/m2);

  8．alcohol or drug abusers within the recent year;

  9．there is a serious heart, lung, kidney, digestive, nervous, mental disease, autoimmune diseases or malignant tumor

  10．drug-induced liver injury;

  11. plan to transplant or have had organ transplants;

  12． are unable or unwilling to provide informed consent or fails to comply with the test requirements;

  13．pregnant, lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-08; Primary Completion 2013-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Efficiency is defined as the patients composition whose ALP level of serum decreased more than 25% compared to baseline at treatment for 24 weeks. | 48 weeks
  After 24 weeks of treatment, calculate the rate of patients whose ALP level of serum ALP decreased more than 25% compared to the baseline. After 48 weeks of treatment, calculate the rate of patients whose ALP level of serum ALP decreased more than 40% compared to the baseline.

SECONDARY OUTCOMES:
The change of laboratory parameters about liver function | 48 weeks
  1. after 24 weeks of treatment, the serum level ALP decreased compared with baseline.
  2. after 24 weeks of treatment, the serum bilirubin level decreased compared with baseline.
  3. after 24 weeks of treatment, the serum level of GGT decreased compared with baseline.
  4. after 24 weeks of treatment, serum ALT, AST levels decreased compared to baseline.
  5. after 48 weeks of treatment, the serum level ALP decreased compared with 24 weeks.
  6. after 48 weeks of treatment, the serum level ALP decreased compared with baseline.
  7. after 48 weeks of treatment, the serum bilirubin level decreased compared with 24 weeks.
  8. after 48 weeks of treatment, the serum level of GGT decreased compared with 24 weeks.
  9. after 48 weeks of treatment, serum ALT, AST levels decreased compared to 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ji Dong Jia, Doctor, Principal Investigator — Beijing Friendship Hospital; Wen Xie, Doctor, Study Director — Beijing Ditan Hospital; Hui Ping Yan, Doctor, Study Director — Beijing YouAn Hospital; Guo Feng Chen, Doctor, Study Director — Beijing 302 Hospital; Gui Qiang Wang, Doctor, Study Director — Peking University First Hospital; Lai Wei, Doctor, Study Director — Peking University People's Hospital; Liu Fang Cheng, Doctor, Study Director — Chinese PLA General Hospital; Min De Zeng, Study Director — RenJi Hospital; Qing Xie, Doctor, Study Director — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine; Guang Feng Shi, Doctor, Study Director — Affiliated HuaShan Hospital of Fudan University; Ji Yao Wang, Doctor, Study Director — Affiliated Zhongshan Hospital of Fudan University; Xiao Hui Miao, Doctor, Study Director — Shanghai Changzheng Hospital; Cheng Wei Chen, Doctor, Study Director — No.85 hospital of PLA; Shan Ming Wu, Doctor, Study Director — Shanghai Public Health Clinical Center; He Ping Hu, Doctor, Study Director — Shanghai Eastern Hepatobiliary Surgery Hospital; Min Hu Chen, Doctor, Study Director — The First Affiliated Hospital,SunYat-Sen University; Zhi Liang Gao, Doctor, Study Director — The Third Affiliated Hospital,SunYat-Sen University; Jin Lin Hou, Doctor, Study Director — Affiliated Southern Hospital of Southern Medical University; Ji Fang Sheng, Doctor, Study Director — The First Affiliated Hospital of Medical College,Zhejiang University; Xiao Qing Fu, Doctor, Study Director — NO.6 People's Hospital of Hangzhou; Hong Tang, Doctor, Study Director — Affiliated Huaxi Hospital of Sichuan University; Ying Han, Doctor, Study Director — The First Affiliated Hospital of the Fourth Military Medical University; Qin Ning, Doctor, Study Director — Affiliated TongJi Hospital Of Tongji Medical College Huazhong University Of Science&Technology; Li Ping Duan, Doctor, Study Director — First Affiliated Hospital of Kunming Medical University; Jie Xu, Doctor, Study Director — NO.3 People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Liver Research Center,Beijing Friendship Hospital, Beijing, Beijing Municipality, China